CLINICAL TRIAL: NCT05426538
Title: Craving to Biologics Used in Severe Asthma
Acronym: CROCUS
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: CROCUS
Record Dates: First submitted 2022-01-05; First posted 2022-06-22 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2021-12

CONDITIONS: Asthma
Keywords: Biological treatment; Patient-reported outcome measures; Treatment evaluation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interview group: A selection of patients will be interviewed, mapping the craving for the next biologic administration. These interviews will be used to develop a questionnaire to quantify the craving for the next administration in the total population.
- Questionnaire group: The remaining patients will be asked to fill in a questionnaire, based on the interviews from Group 1.

SUMMARY:
Some patients treated with biologics for severe asthma experience a craving to the next biological administration. This phenomenon has never been described before. In this study, the researchers aim to further elucidate the feeling of needing the next administration of a biologic for severe asthma.

DETAILED DESCRIPTION:
Recent research by Kroes and colleagues on omalizumab levels has shown that approximately half of patients on long-term omalizumab therapy (>4 months) experience a subjective craving for the next dose. These patients had a need (Borg scale 3-10) for the next dose of biologic before the usual periodic dose, while other patients indicated that they had no or a low need (Borg scale 0-2) for the next dose at the usual dosing moment. This so-called 'craving' has not been described in the literature before. Patients in the high-requirement group had significantly lower median omalizumab trough levels than patients in the low-requirement group. There may be a relationship between blood levels of biologics and the need for the next dose. However, data is currently only available on the variability in serum trough levels of omalizumab, but not yet on the other biologics for asthma, some of which are administered as a fixed dose and some are dosed by body weight. No assays are currently available for blood level determinations from the other biologics.

Before investigating the relationship between blood levels and the need for biologics, it is important to fully map the 'craving'. Some patients who are responders to biologic therapy based on improvements in clinical outcomes still do not have good enough control of their asthma and indicate that the dosing interval is not optimal. In addition to patients that indicate a need for the next dose, there are also patients that would like a longer dosing interval. To date, dosing interval adjustments have been made based on the patient's subjective experience and the physician's clinical judgment. This study investigates how big the problem of need for the next dose is, how patients experience this need, what this need exactly entails, whether this occurs more often in patients treated for a longer period and what possible problems patients experience in the treatment with biologics against serious problems.

ELIGIBILITY:
Inclusion Criteria:

* Treated with a biologic for severe asthma in the Medical Centre Leeuwarden for more than 4 months

Exclusion Criteria:

* Not speaking Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population concerns patients in the Medical Center Leeuwarden (MCL) with severe asthma who are treated with a biologic (omalizumab, mepolizumab, reslizumab, benralizumab or dupilumab) for more than 4 months.
  A treatment duration longer than 4 months has been chosen, so that only responders to the biologics are included in the study and the therapy has its effect.
  About 20 patients are interviewed. Subsequently, the questionnaire will be presented to approximately 30 patients per biologic, a total of approximately 150 patients.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of craving to the next biologic administration. | 6 months
  Craving will be assessed as a BORG-scale score >2. This scale ranges from 0 (No craving at all) to 10 (Extreme craving).
The character of craving to the next biologic administration. | 6 months
  This will be assessed by scoring the prevalence of asthma-related symptoms in patients reporting a craving. Craving will be assessed as a BORG-scale score >2. This scale ranges from 0 (No craving at all) to 10 (Extreme craving).

SECONDARY OUTCOMES:
Differences in craving (BORG-scale 0-10) between patients treated for more or less than 1 year. | 6 months
  Craving will be assessed with a BORG-scale score. This scale ranges from 0 (No craving at all) to 10 (Extreme craving).
Differences in craving (BORG-scale 0-10) between patients with different biologics. | 6 months
  Craving will be assessed with a BORG-scale score. This scale ranges from 0 (No craving at all) to 10 (Extreme craving).
Any other issues regarding the craving/administration of biologics for severe asthma, based on patient-level input from interviews. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Provincie Friesland, Netherlands

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared, since data is collected in private interviews.